CLINICAL TRIAL: NCT02666105
Title: Phase II Trial of Exemestane in Previously Treated Post-Menopausal Women With Advanced Non-Small Cell Lung Cancer
Brief Title: Exemestane in Post-Menopausal Women With NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015LS095
Record Dates: First submitted 2016-01-22; First posted 2016-01-28 (Estimated); Results first posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Exemestane Therapy (Experimental)
  Interventions: Drug: Exemestane

INTERVENTIONS:
Drug: Exemestane — One 25 mg tablet once daily for a minimum of 6 weeks
  Other Names: Aromasin

SUMMARY:
This is a phase II therapeutic study of adding exemestane therapy in post-menopausal women with advanced non-small cell lung cancer (NSCLC) who are progressing while on treatment with an immune checkpoint antibody (pembrolizumab, atezolizumab, or nivolumab).

ELIGIBILITY:
Inclusion Criteria

* Recurrent or progressive advanced stage non-small cell lung cancer (no small cell component) with most recent treatment being an FDA approved immune checkpoint inhibitor (pembrolizumab, atezolizumab, or nivolumab) NOTE: Pathology reports documenting the diagnosis of NSCLC are required to be reviewed to confirm outside diagnosis
* Sufficient tumor tissue available from original diagnosis or subsequent biopsy for analysis of estrogen receptor and aromatase - tumor block or a minimum of 5 unstained slides
* Failed at least 1 prior FDA approved treatment for advanced NSCLC. Patients with EGFR/ALK/ROS1 rearrangements should have received an FDA-approved TKI prior to enrollment on this trial.
* Measureable disease by RECIST version 1.1
* Post-menopausal defined as

  * Age ≥ 55 years and 1 year or more of amenorrhea
  * Age < 55 years and 1 year or more of amenorrhea with an estradiol assay < 20 pg/mL
  * Surgical menopause with bilateral oophorectomy
* ECOG performance status 0, 1 or 2

  * Life expectancy of 3 months or more in the opinion of the enrolling investigator and documented in the medical record
* Adequate organ function within 14 days of study enrollment defined as:

  * Hematology:

    ** Absolute neutrophil count (ANC) ≥ 1500/mm³, Platelets ≥ 100,000/mm³, Hemoglobin ≥ 8 g/dL
  * Biochemistry:

    * Total Bilirubin within normal institutional limits
    * AST/SGOT and ALT/SGPT ≤ 2.5 x upper limit of normal (ULN), except if there is known hepatic metastasis, wherein transaminases may be ≤ 5 x institutional ULN.
    * Serum creatinine ≤ 1.5 mg/dl or glomerular filtration rate > 50 ml/min
* Must have recovered to CTCAE v 4 Grade 1 or better from the acute effects of any prior surgery, chemotherapy or radiation therapy. Chronic residual toxicity (i.e. peripheral neuropathy) is permitted.
* A minimum time period must elapse between the end of a previous treatment and start of study therapy:

  * 1 week from the completion of radiation therapy for brain metastases
  * 4 weeks from the completion of chemotherapy or any experimental therapy
  * 4 weeks from prior major surgery (such as open biopsy or significant traumatic injury)
* Voluntary written consent before any research related procedures or therapy

Exclusion Criteria

* Known active CNS disease - If patient has history of brain metastases, the brain lesions must have been treated with radiation and/or surgery - patients should be neurologically stable and requiring ≤10mg oral prednisone equivalence of steroids per day
* Any toxicity from immune-related toxicity from prior immune therapy that would preclude further treatment with anti-PD-1/PDL-1 inhibitor or ongoing IR toxicity ≥ Grade 2
* Requiring > 10 mg prednisone equivalence of steroids per day for immune-related toxicity
* Inability or unwilling to swallow study drug
* Any gastrointestinal condition causing malabsorption or obstruction (eg, celiac sprue, gastric bypass surgery, strictures, adhesions, history of small bowel resection, blind loop syndrome)
* Currently using hormone replacement therapy (oral or patch) or/and phytoestrogen supplements (i.e. black cohosh)
* Known hypersensitivity to exemestane or its excipients
* Any serious underlying medical condition that, in the opinion of the enrolling physician, would impair the ability of the patient to receive protocol treatment
* Prior malignancy, with the exception of curatively treated squamous cell or basal carcinoma of the skin or in situ cervical cancer, unless there is a 3-year disease-free interval
* Concomitant use of strong CYP3A4 inducers such as rifampicin, phenytoin, carbamazepine, phenobarbital, or St. John's wort as these may significantly reduce the availability of exemestane

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manish Patel, DO, Principal Investigator — University of Minnesota Masonic Cancer Center
Locations (18):
- United States (18):
  - Mayo Clinic Health System, Albert Lea, Minnesota
  - Essentia Health St. Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health Deer River, Deer River, Minnesota
  - Essentia Health St. Mary's Detroit Lakes, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Fosston, Fosston, Minnesota
  - Fairview Grand Itasca Clinic & Hospital, Grand Rapids, Minnesota
  - Essentia Health Hibbing, Hibbing, Minnesota
  - Fairview Range Medical Center, Hibbing, Minnesota
  - Mayo Clinic Health System, Mankato, Minnesota
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Monticello Cancer Center (MMCORC), Monticello, Minnesota
  - Essentia Health Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia, Virginia, Minnesota
  - Sanford Worthington Medical Center, Worthington, Minnesota

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exemestane Therapy
Started | 6
Completed | 5
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Post-Menopausal Women
Arm/Group | Exemestane Therapy
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Disease Response (RECIST)
Description: Initial disease response will be assessed from 6 weeks to 1 year after the start of exemestane using the Response Criteria in Solid Tumors (RECIST). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 6 weeks
Measure: Mean (Full Range); unit: days
Arm/Group | Exemestane Therapy
Number analyzed (Participants) | 6
days | NA [NA to NA] — Insufficient number of participants with events.

2. Secondary Outcome: Toxicity Assessment
Description: Toxicity will be assessed from the 1st dose to Post Treatment Day 30, up to 22 weeks. Toxicity severity will be graded using the Common Toxicity Criteria for Adverse Events (CTCAE) version 4.
Time Frame: Post Treatment Day 30
Measure: Number; unit: Adverse Events
Arm/Group | Exemestane Therapy
Number analyzed (Participants) | 5
Adverse Events | 14

3. Secondary Outcome: Progression-free Survival
Description: progression-free survival will be assessed until 1 year after study enrollment based on the definitions found in RECIST 1.1
Time Frame: 1 year after enrollment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Exemestane Therapy
Number analyzed (Participants) | 6
Percentage of participants | 17 [1 to 52]

4. Secondary Outcome: Quality of Life Assessment
Description: Quality of life will be assessed by use of Patient-Reported Outcomes Measurement Information System 29 (PROMIS-29) at baseline, every 3 weeks from the 1st dose to Post Treatment Day 30, up to 22 weeks. Patient's report on a number of subjects on a 0-10 scale. The scores range from 28 to 150. 50 is the average score, 28 is the best health and 150 is the worst health.
Time Frame: Baseline, Treatment, End of Treatment, and 1 Month Post-Treatment
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Groups:
- Exemestane Therapy - Baseline: Quality of life assessment at baseline.
- Exemestane Therapy - 3 Weeks: Quality of life assessment at three weeks of treatment.
- Exemestane Therapy - 6 Weeks: Quality of life assessment at six weeks of treatment.
- Exemestane Therapy - 9 Weeks: Quality of life assessment at nine weeks of treatment.
- Exemestane Therapy - 12 Weeks: Quality of life assessment at twelve weeks of treatment.
- Exemestane Therapy - 15 Weeks: Quality of life assessment at fifteen weeks of treatment.
- Exemestane Therapy - 18 Weeks: Quality of life assessment at end of treatment, eighteen weeks of treatment.
- Exemestane Therapy - 1 Month Post-Treatment: Quality of life assessment one month post-treatment.
Arm/Group | Exemestane Therapy - Baseline | Exemestane Therapy - 3 Weeks | Exemestane Therapy - 6 Weeks | Exemestane Therapy - 9 Weeks | Exemestane Therapy - 12 Weeks | Exemestane Therapy - 15 Weeks | Exemestane Therapy - 18 Weeks | Exemestane Therapy - 1 Month Post-Treatment
Number analyzed (Participants) | 4 | 4 | 3 | 3 | 2 | 2 | 2 | 2
Score on a scale | 44 [44 to 45] | 52 [41 to 88] | 45 [41 to 57] | 51 [48 to 115] | 46 [40 to 51] | 57 [46 to 67] | 55 [41 to 69] | 57 [46 to 68]

ADVERSE EVENTS:
Time Frame: Monitoring for adverse events will begin with the start of the exemestane and continue through and including 28 calendar days after the last dose of exemestane, an average of 22 weeks.
Arm/Group | Exemestane Therapy
All-Cause Mortality (participants affected / at risk) | 3/6
Serious Adverse Events (participants affected / at risk) | 6/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exemestane Therapy (N=6)
Dehydration (Metabolism and nutrition disorders) | 1 (1) — Grade 3
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 5
Sepsis (Infections and infestations) | 1 (1) — Grade 4
Skin infection (Infections and infestations) | 1 (1) — Grade 3
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) — Grade 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Grade 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Exemestane Therapy (N=6)
Edema limbs (General disorders) | 3/5 (3)
Pain (General disorders) | 2/5 (2)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1/5 (1)
Weight gain (Investigations) | 1/5 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2/5 (2)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1/5 (1)
Anemia (Blood and lymphatic system disorders) | 3/5 (11)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1/5 (1)
Eye disorders - Other, specify (Eye disorders) | 1/5 (1)
Abdominal pain (Gastrointestinal disorders) | 1/5 (1)
Diarrhea (Gastrointestinal disorders) | 1/5 (2)
Fatigue (General disorders) | 1/5 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1/5 (1)
Immune system disorders - Other, specify (Immune system disorders) | 1/5 (2)
Sepsis (Infections and infestations) | 1/5 (1)
Upper respiratory infection (Infections and infestations) | 2/5 (2)
Urinary tract infection (Infections and infestations) | 1/5 (1)
Alanine aminotransferase increased (Investigations) | 1/5 (15)
Alkaline phosphatase increased (Investigations) | 1/5 (5)
Aspartate aminotransferase increased (Investigations) | 1/5 (8)
Blood bilirubin increased (Investigations) | 1/5 (2)
Cardiac troponin I increased (Investigations) | 1/5 (1)
Lymphocyte count decreased (Investigations) | 1/5 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1/5 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1/5 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1/5 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1/5 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1/5 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1/5 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2/5 (2)
Hot flashes (Vascular disorders) | 1/5 (1)
Lymphedema (Vascular disorders) | 1/5 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/05/NCT02666105/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT02666105/ICF_001.pdf